CLINICAL TRIAL: NCT02987946
Title: Optimizing Anti Coagulant Therapy in Neurosurgical Interventions in Patients with an Increased Risk for Thrombo-embolic Complications
Brief Title: Leiden Trial in Prevention of Post-Operative ThromboEmbolic Events
Acronym: TIPOTEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, C.L.A.Vleggeert-Lankamp, MD MSc PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL56552.058.16
Record Dates: First submitted 2016-11-16; First posted 2016-12-09 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2024-06

CONDITIONS: Deep-Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Nadroparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fraxiparine (Active Comparator): Intervention: All patients receive Fraxiparine 2850 IE daily, starting preoperatively compatible with current practice. After randomization the patients in this arm will be subjected to fraxipareine 2850 IE daily. According to current guidelines in the LUMC the Fraxiparine dose is doubled to 5600 IE in patients with a weight above 100 kg.
  Interventions: Drug: Fraxiparine
- IPD (Experimental): Intervention: IPD Device: After randomization the patients in this arm will be subjected to fraxiparine 2850 IE daily and intermittent pressure devices for at least 48 hours or until mobilization. The intermittent pressure device is a leg pump delivered by Converis(R).
  Interventions: Device: IPD Device delivered by Converis; Drug: Fraxiparine

INTERVENTIONS:
Device: IPD Device delivered by Converis — After randomization patients will be subjected to perioperative (48 hrs) intermittent pneumatic compression.
  Other Names: IPD
  Arms: IPD
Drug: Fraxiparine — All patients receive Fraxiparine 2850 IE daily, starting preoperatively compatible with current practice.
  Other Names: LMWH

SUMMARY:
In neurosurgical patients, the risk for venous thromboembolic events (VTE) is high due to the relatively long duration of surgery, the high occurrence of prolonged immobilization of patients due to paresis of the legs or intracranial pathology causing inability to mobilise2. Moreover, intracranial and intraspinal tumours and subarachnoid haemorrhage cause hypercoagulability, which increases the risk on VTE. There is a high degree of diversity in attributed risk on thrombosis in the neurosurgical patient cohort. Due to this diversity, insufficient power of performed studies and lack of careful phenotyping and description of risk factors in previous studies on deep venous thrombosis (DVT) prophylaxis, as yet the optimal DVT prophylaxis in neurosurgery remains unclear. A prospective randomized study with adequate power and detailed information on patient related factors (malignancy, subarachnoid haemorrhage, prevailing coagulopathies), type of surgery, duration of surgery, and postoperative immobilisation will allow us to identify the optimal treatment strategy for high risk neurosurgical patients.

In the current study all patients that fulfil the inclusion criteria will be subjected to post-operative systematic evaluation of VTE by echo-duplex investigation.

DETAILED DESCRIPTION:
It is clear that thrombo-embolic prophylaxis is mandatory in neurosurgical interventions. The current prophylactic strategy using preoperatively started low molecular-weight heparine (LMWH) allows still a considerable number of thrombo-embolic complications, in particular in those patients that are subjected to prolonged neurosurgical interventions. Guidelines advise mechanical prophylaxis. However, these guidelines are based on literature with low grade of evidence. To achieve the highest grade of evidence we will randomize subsequent patients between intermittent compression stockings with preoperative LMWH prophylaxis, and LMWH as stand alone prophylaxis. The last, being the current state of practice in all neurosurgical patients in our ward, including the high thrombosis risk group. All patients will receive preoperatively started LMWH.

There is a high degree of diversity in attributed risk on thrombosis in the neurosurgical patient cohort. Due to this diversity, insufficient power of performed studies and lack of careful phenotyping and description of risk factors in previous studies on deep venous thrombosis (DVT) prophylaxis, as yet the optimal DVT prophylaxis in neurosurgery remains unclear. A prospective randomized study with adequate power and detailed information on patient related factors (malignancy, subarachnoid haemorrhage, prevailing coagulopathies), type of surgery, duration of surgery, and postoperative immobilisation will allow us to identify the optimal treatment strategy for high risk neurosurgical patients.

In the current study all patients that fulfil the inclusion criteria will be subjected to post-operative systematic evaluation of venous thromboembolic events (VTE) by echo-duplex investigation.

• 2. Goal of the study The primary goal of the current study is to investigate whether the combination of perioperative intermittent pneumatic compression and LMWH has a lower incidence of postoperative thrombo-embolic complications within a week after a high risk neurosurgical intervention in comparison to patients receiving merely LMWH prophylaxis.

Secondary research questions are:

* Is there a difference in number of patients with clinical symptoms of thromboembolus in patients receiving the combination of peroperative intermittent pneumatic compression of the lower limbs and LMWH in comparison to patients receiving merely LMWH prophylaxis in high risk neurosurgical patients, scored two months after surgery;
* What is the prevalence of VTE in high risk neurosurgical patients in the Leiden University Medical Centre (LUMC) receiving LMWH prophylaxis;
* What are the risk factors for the prevalence of VTE in high risk neurosurgical patients in the LUMC;
* What is the incidence of bleeding complications in high risk neurosurgical patients in the LUMC receiving LMWH prophylaxis;
* Is there a difference in length of hospital stay in patients receiving the combination of peroperative intermittent pneumatic compression of the lower limbs and LMWH in comparison to patients receiving merely LMWH prophylaxis in high risk neurosurgical patients;
* Is there a difference in patient perceived recovery at discharge and at 2 month follow up in patients receiving the combination of perioperative intermittent pneumatic compression and LMWH in comparison to patients receiving merely LMWH prophylaxis in high risk neurosurgical patients;
* Is there a difference in Quality of life at discharge and at 2 month follow up in patients receiving the combination of perioperative intermittent pneumatic compression of the legs and LMWH in comparison to patients receiving merely LMWH prophylaxis in high-risk neurosurgical patients;
* Is it relevant to consider cost-effectiveness of the use of perioperative intermittent pneumatic compression of the legs and if so, what is the cost-effectiveness?
* 3. Randomized controlled trial This is a randomized controlled trial on high-risk neurosurgical patients in a University hospital (see inclusion and exclusion criteria) in which consecutive patients who meet the inclusion criteria are invited to participate in the trial. Clinical and demographic data are gathered, as well as surgical details and prevailing complications. Postoperative bleeding requiring secondary surgery or lengthening of hospital stay will be documented as a clinically relevant bleeding complication. All patients receive Fraxiparine 2850 IU (international units) daily, starting preoperatively compatible with current practice. At admission patients will be randomized to be subjected to perioperative (48 hrs) intermittent pneumatic compression or standard care. Following current guidelines in the LUMC the Fraxiparine dose is doubled to 5600 IU in patients with a weight above 100 kg.

All randomized patients will receive a postoperative doppler examination of the major veins of both lower limb in order to identify a possible VTE. A post-operative thrombo-embolic complication is defined as follows7:

1. Asymptomatic VTE confirmed by echo Doppler;
2. Symptomatic VTE confirmed by echo Doppler;
3. Symptomatic pulmonary embolism (PE) confirmed by CT scan
4. Fatal pulmonary embolism confirmed by autopsy

> 3.1 Population The neurosurgical patient has an increased risk on thrombo-embolic complications because he is subjected to an intervention that in general takes a long time and causes the patient to be immobilized during a longer period (during and directly after surgery). Moreover, the pathology is frequently carcinomatous, having an increased risk for thrombo-embolic events by nature. The in- and exclusion criteria are aiming at these properties of the patients. All consecutive patients that fulfil the criteria will be invited to participate in this study. In order to be included the patient has to sign an informed consent. Based on a power analysis 140 patients in both randomization arms have to be included (based on a VTE incidence of 15% which will decrease to 5% after treatment with intermittent pneumatic leg pumps during surgery; alpha 0.05, power 80%) to be able to obtain a significant effect.

ELIGIBILITY:
Inclusion Criteria:• Intracranial surgery;

* Tumour surgery (spinal or intracranial);
* >180 min estimated surgical intervention time;
* >240 min time under anaesthesia;
* Spine trauma surgery;

Exclusion Criteria:

* • Age under 18 years;

  * Perioperative continuation of anti coagulant therapy indicated other than prophylactic LMWH;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Lower incidence of thromboembolic complications in patients with IPD + LMWH by adding IPD to usual care, established with systematic doppler/duplex evaluation in all patients at 5 +/- 2 days post surgery | 1 week
  The primary goal of the current study is to investigate whether the combination of perioperative intermittent pneumatic compression and LMWH has a lower incidence of postoperative thrombo-embolic complications within a week after a high risk neurosurgical intervention in comparison to patients receiving merely LMWH prophylaxis. All patients will be subjected to doppler/duplex in the week after surgery. Follow up of all patients will be performed at 5 +/- 2 days after surgery, during admission time. At this time all patient will have a duplex ultrasound examination to assess the prevalence of a possible deep venous thrombosis. This period has been chosen in analogy with existing literature (appendix A). 9-15 For this examination patients have to be able stand upright. Therefore in some cases (e.g ICU patients) the interval will be longer, with a maximum of 20 days.

SECONDARY OUTCOMES:
prevalence of DVT measured by duplex/doppler routinely performed in the whole study population | 1 week
Clinical signs of DVT i.e. swollen,painful and red leg or pulmonary embolism | 2 months
Quality of life by EQ-5D | 2 mos after surgery
Patient perceived recovery with Likert scale | 2 months
Cost effectiveness with EQ-5D and estimated costs in cost diaries | 2 months
  is the additional use of IPD cost effective in prevention of DVT in neurosurgical patients

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Vleggeert-Lankamp, MD MSc PhD, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided